CLINICAL TRIAL: NCT00976937
Title: A Randomized, Double-blind, Double-dummy, 2-arm Parallel-group, Multicenter 24-week Study Comparing the Efficacy and Safety of AVE0010 to Sitagliptin as add-on to Metformin in Obese Type 2 Diabetic Patients Younger Than 50 and Not Adequately Controlled With Metformin
Brief Title: 24-week Study Comparing Lixisenatide to Sitagliptin as add-on to Metformin in Obese Type 2 Diabetic Patients Younger Than 50 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC10780; EudraCT:2008-007 334-22
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lixisenatide (Experimental): 2-step initiation regimen of lixisenatide along with sitagliptin placebo: lixisenatide 10 microgram (mcg) once daily (QD) for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24 along with placebo matching to sitagliptin 100 milligram (mg) capsule orally QD up to Week 24.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector; Drug: Sitagliptin Placebo; Drug: Metformin
- Sitagliptin (Active Comparator): Sitagliptin along with 2-step initiation regimen of volume matching lixisenatide placebo: sitagliptin 100 mg capsule orally QD up to Week 24 along with volume matching lixisenatide placebo 10 mcg QD for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24.
  Interventions: Drug: Lixisenatide Placebo; Device: Pen auto-injector; Drug: Sitagliptin; Drug: Metformin

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Self-administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Lixisenatide
Drug: Lixisenatide Placebo — Self-administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Sitagliptin
Device: Pen auto-injector
  Other Names: OptiClik®
Drug: Sitagliptin — Administered orally once a day in the morning with or without food at approximately the same time each day.
  Other Names: Januvia®
  Arms: Sitagliptin
Drug: Sitagliptin Placebo — Administered orally once a day in the morning with or without food at approximately the same time each day.
  Arms: Lixisenatide
Drug: Metformin — Metformin to be continued at stable dose (at least 1.5 gram per day) up to Week 24.

SUMMARY:
The purpose of this study is to evaluate benefits and risks of lixisenatide (AVE0010), in comparison to sitagliptin, as an add-on treatment to metformin, in obese (body mass index [BMI] greater than or equal to 30 kilogram per square meter [kg/m^2]) type 2 diabetic patients less than 50 years of age, over a period of 24 weeks of treatment.

The primary objective of this study is to assess the efficacy of lixisenatide, in comparison to sitagliptin, as an add-on treatment to metformin on a composite endpoint of glycemic control in terms of glycosylated hemoglobin (HbA1c) and body weight, at Week 24.

Secondary objectives are to assess the effects of lixisenatide, in comparison to sitagliptin, as an add-on treatment to metformin on absolute changes in HbA1c values and body weight; fasting plasma glucose (FPG); plasma glucose, insulin, C-peptide, glucagon, and proinsulin during a 2-hour standardized meal test; insulin resistance assessed by homeostatic model assessment of insulin resistance (HOMA-IR); beta cell function assessed by homeostatic model assessment of beta-cell function (HOMA-beta); to evaluate safety, tolerability, and anti-lixisenatide antibody development.

ELIGIBILITY:
Inclusion criteria

* Type 2 diabetes mellitus, diagnosed for at least 1 year at the time of screening visit, insufficiently controlled with metformin at a stable dose of at least 1.5 gram/day (g/day) for at least 3 months prior to the screening visit
* Patients with obesity (BMI greater than equal to [>=] 30 kg/m^2) and aged from 18 years to less than 50 years

Exclusion criteria

* HbA1c less than (<) 7.0 percent (%) or HbA1c greater than (>) 10% at screening
* Type 1 diabetes mellitus
* Pregnant or breastfeeding women or women of childbearing potential with no effective contraceptive method
* FPG at screening >250 milligram/deciliter (mg/dL) (>13.9 millimole/ liter [mmol/L])
* Weight change of more than 5 kg during the 3 months preceding the screening visit
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease, personal or family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC (for example, multiple endocrine neoplasia syndromes)
* History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening
* Hemoglobinopathy or hemolytic anemia or receipt of blood or plasma products within 3 months prior to the time of screening
* Within the last 6 months prior to screening: history of myocardial infarction, stroke, or heart failure requiring hospitalization
* Known history of drug or alcohol abuse within 6 months prior to the time of screening
* Any clinically significant abnormality identified on physical examination, laboratory tests, electrocardiogram (ECG) or vital signs at the time of screening that in the judgment of the investigator or any sub-investigator could have precludes safe completion of the study or constrains efficacy assessment such as major systemic diseases, presence of clinically significant diabetic retinopathy or presence of macular edema likely to require laser treatment within the study period
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting systolic or diastolic blood pressure >180 millimeter of mercury (mmHg) or >110 mmHg, respectively
* Laboratory findings at the time of screening : Amylase and/or lipase >3 times the upper limit of normal (ULN) laboratory range; alanine aminotransferase (ALT): >3 times ULN; total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome); hemoglobin <11 gram/deciliter and/or neutrophils <1500 per cubic millimeter (mm^3) and/or platelets <100 000/mm^3; positive test for Hepatitis B surface antigen (HBsAg) and/or Hepatitis C antibody (HCAb), positive serum pregnancy test in females of childbearing potential, and calcitonin >=20 picogram per milliliter (pg/mL) (5.9 picomole per liter)
* Patients who are considered by the investigator or any sub-investigator as inappropriate for the study for any reason (for example, impossibility to meet specific protocol requirements [such as scheduled visits, being able to do self-injections], likelihood of requiring treatment during the screening phase and treatment phase with drugs not permitted by the clinical study protocol, investigator or any sub-investigator, pharmacist, study coordinator, other study staff or relative thereof directly involved in the conduct of the protocol)
* Use of other oral or injectable antidiabetic or hypoglycemic agents than metformin (for example, sulfonylurea, alpha glucosidase inhibitor, thiazolidinedione, exenatide, dipeptidyl peptidase IV (DPP-IV) inhibitors, insulin) within 3 months prior to the time of screening
* History of bariatric surgery, anti-obesity treatment, or unstable diet within 3 months prior to the time of screening
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for one week or more within 3 months prior to the time of screening
* Use of any investigational drug within 3 months prior to screening
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including (but not limited to): gastroparesis, unstable (that is, worsening) and not controlled (that is, prolonged nausea and vomiting) gastroesophageal reflux disease requiring medical treatment, within 6 months prior to the time of screening
* Any previous treatment with lixisenatide (for example, participation in a previous study with lixisenatide)
* Allergic reaction to any glucagon like peptide-1 (GLP 1) agonist in the past (for example, exenatide, liraglutide) or to metacresol
* History of a serious hypersensitivity reaction to sitagliptin
* Moderate or severe renal impairment (creatinine clearance inferior to 50 milliliter/minute [mL/min])
* Additional exclusion criteria at the end of the run-in phase: informed consent withdrawal; lack of compliance during the single-blind placebo run-in period (>2 injections missed or >2 capsules missed); and patient with any adverse event which could have precludes the inclusion in the study, as assessed by the investigator

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 319 (Actual)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (92):
- United States (21):
  - Sanofi-Aventis Investigational Site Number 840019, Montgomery, Alabama
  - Sanofi-Aventis Investigational Site Number 840003, Muscle Shoals, Alabama
  - Sanofi-Aventis Investigational Site Number 840022, Mesa, Arizona
  - Sanofi-Aventis Investigational Site Number 840011, Anaheim, California
  - Sanofi-Aventis Investigational Site Number 840014, Paramount, California
  - Sanofi-Aventis Investigational Site Number 840027, Redlands, California
  - Sanofi-Aventis Investigational Site Number 840021, Augusta, Georgia
  - Sanofi-Aventis Investigational Site Number 840007, Roswell, Georgia
  - Sanofi-Aventis Investigational Site Number 840016, Chicago, Illinois
  - Sanofi-Aventis Investigational Site Number 840018, Chicago, Illinois
  - Sanofi-Aventis Investigational Site Number 840001, Evansville, Indiana
  - Sanofi-Aventis Investigational Site Number 840002, Baton Rouge, Louisiana
  - Sanofi-Aventis Investigational Site Number 840031, Clarkston, Michigan
  - Sanofi-Aventis Investigational Site Number 840020, Florissant, Missouri
  - Sanofi-Aventis Investigational Site Number 840006, Butte, Montana
  - Sanofi-Aventis Investigational Site Number 840026, Perrysburg, Ohio
  - Sanofi-Aventis Investigational Site Number 840004, Medford, Oregon
  - Sanofi-Aventis Investigational Site Number 840025, Altoona, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840009, Brentwood, Tennessee
  - Sanofi-Aventis Investigational Site Number 840008, Dallas, Texas
  - Sanofi-Aventis Investigational Site Number 840010, San Antonio, Texas
- Australia (6):
  - Sanofi-Aventis Investigational Site Number 036006, Adelaide
  - Sanofi-Aventis Investigational Site Number 036001, Box Hill
  - Sanofi-Aventis Investigational Site Number 036004, Elizabeth Vale
  - Sanofi-Aventis Investigational Site Number 036002, Geelong
  - Sanofi-Aventis Investigational Site Number 036005, Meadowbrook
  - Sanofi-Aventis Investigational Site Number 036003, Sydney
- Brazil (7):
  - Sanofi-Aventis Investigational Site Number 076005, Belém
  - Sanofi-Aventis Investigational Site Number 076001, Brasília
  - Sanofi-Aventis Investigational Site Number 076006, Caxias do Sul
  - Sanofi-Aventis Investigational Site Number 076003, Curitiba
  - Sanofi-Aventis Investigational Site Number 076002, Rio de Janeiro
  - Sanofi-Aventis Investigational Site Number 076004, São Paulo
  - Sanofi-Aventis Investigational Site Number 076007, São Paulo
- Canada (10):
  - Sanofi-Aventis Investigational Site Number 124004, Calgary
  - Sanofi-Aventis Investigational Site Number 124008, Hamilton
  - Sanofi-Aventis Investigational Site Number 124005, London
  - Sanofi-Aventis Investigational Site Number 124006, Montreal
  - Sanofi-Aventis Investigational Site Number 124013, Oakville
  - Sanofi-Aventis Investigational Site Number 124002, Saint Romuald
  - Sanofi-Aventis Investigational Site Number 124012, Thornhill
  - Sanofi-Aventis Investigational Site Number 124011, Toronto
  - Sanofi-Aventis Investigational Site Number 124003, Vancouver
  - Sanofi-Aventis Investigational Site Number 124007, Victoria
- Chile (5):
  - Sanofi-Aventis Investigational Site Number 152001, Santiago
  - Sanofi-Aventis Investigational Site Number 152004, Santiago
  - Sanofi-Aventis Investigational Site Number 152003, Santiago
  - Sanofi-Aventis Investigational Site Number 152002, Santiago
  - Sanofi-Aventis Investigational Site Number 152005, Santiago
- Germany (3):
  - Sanofi-Aventis Investigational Site Number 276002, Berlin
  - Sanofi-Aventis Investigational Site Number 276005, Ludwigshafen
  - Sanofi-Aventis Investigational Site Number 276004, Schkeuditz
- Guatemala (5):
  - Sanofi-Aventis Investigational Site Number 320002, Guatemala City
  - Sanofi-Aventis Investigational Site Number 320001, Guatemala City
  - Sanofi-Aventis Investigational Site Number 320004, Guatemala City
  - Sanofi-Aventis Investigational Site Number 320005, Guatemala City
  - Sanofi-Aventis Investigational Site Number 320006, Guatemala City
- Mexico (10):
  - Sanofi-Aventis Investigational Site Number 484003, Aguascalientes
  - Sanofi-Aventis Investigational Site Number 484010, Chihuahua City
  - Sanofi-Aventis Investigational Site Number 484009, Chihuahua City
  - Sanofi-Aventis Investigational Site Number 484012, Df
  - Sanofi-Aventis Investigational Site Number 484008, Mérida
  - Sanofi-Aventis Investigational Site Number 484011, México
  - Sanofi-Aventis Investigational Site Number 484001, Pachuca
  - Sanofi-Aventis Investigational Site Number 484005, Pachuca
  - Sanofi-Aventis Investigational Site Number 484006, Veracruz
  - Sanofi-Aventis Investigational Site Number 484002, Zapopan
- Peru (5):
  - Sanofi-Aventis Investigational Site Number 604005, Lima
  - Sanofi-Aventis Investigational Site Number 604003, Lima
  - Sanofi-Aventis Investigational Site Number 604001, Lima
  - Sanofi-Aventis Investigational Site Number 604002, Lima
  - Sanofi-Aventis Investigational Site Number 604004, Lima
- Poland (4):
  - Sanofi-Aventis Investigational Site Number 616002, Bialystok
  - Sanofi-Aventis Investigational Site Number 616001, Bydgoszcz
  - Sanofi-Aventis Investigational Site Number 616006, Warsaw
  - Sanofi-Aventis Investigational Site Number 616003, Wroclaw
- Romania (8):
  - Sanofi-Aventis Investigational Site Number 642004, Bacau
  - Sanofi-Aventis Investigational Site Number 642006, Bucharest
  - Sanofi-Aventis Investigational Site Number 642008, Bucharest
  - Sanofi-Aventis Investigational Site Number 642010, Iași
  - Sanofi-Aventis Investigational Site Number 642009, Ploieşti
  - Sanofi-Aventis Investigational Site Number 642001, Reşiţa
  - Sanofi-Aventis Investigational Site Number 642005, Suceava
  - Sanofi-Aventis Investigational Site Number 642007, Timișoara
- Russia (5):
  - Sanofi-Aventis Investigational Site Number 643002, Kazan'
  - Sanofi-Aventis Investigational Site Number 643001, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643003, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643005, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643004, Tyumen
- Ukraine (3):
  - Sanofi-Aventis Investigational Site Number 804003, Chernivtsi
  - Sanofi-Aventis Investigational Site Number 804001, Kiev
  - Sanofi-Aventis Investigational Site Number 804004, Kyiv

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 92 centers in 13 countries between August 31, 2009 and March 19, 2011.
Pre-assignment Details: A total of 620 patients were screened of which 301 (48.5%) were screen failures; main reason for screen failure was glycosylated hemoglobin (HbA1c) values being out of the defined protocol range (greater than or equal to 7% and less than or equal to 10%). A total of 319 patients were randomized.
Groups:
- Lixisenatide: 2-step initiation regimen of lixisenatide along with sitagliptin placebo: lixisenatide 10 microgram (mcg) once daily (QD) subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24 along with placebo matching to sitagliptin 100 milligram (mg) capsule orally QD up to Week 24.
- Sitagliptin: Sitagliptin along with 2-step initiation regimen of volume matching lixisenatide placebo: sitagliptin 100 mg capsule orally QD up to Week 24 along with volume matching lixisenatide placebo 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24.
Period: Overall Study
Arm/Group | Lixisenatide | Sitagliptin
Started | 158 (Randomized) | 161
Treated/Safety Population | 158 (All patients who were exposed to at least 1 dose, regardless of amount of treatment administered.) | 161
Modified Intent-to-Treat(mITT)Population | 158 (All randomized patients who received at least 1 dose of study drug.) | 161
Completed | 142 | 150
Not Completed | 16 | 11
Not completed — Adverse Event | 4 | 5
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Poor compliance to protocol | 3 | 0
Not completed — Personal and Familial Reason | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Lixisenatide: 2-step initiation regimen of lixisenatide along with sitagliptin placebo: lixisenatide 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24 along with placebo matching to sitagliptin 100 mg capsule orally QD up to Week 24.
- Total: Total of all reporting groups
Arm/Group | Lixisenatide | Sitagliptin | Total
Number analyzed (Participants) | 158 | 161 | 319
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (5.2) | 43.4 (4.7) | 43.1 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 88 | 191
  Male | 55 | 73 | 128
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Caucasian/White | 132 | 127 | 259
  Race: Black | 8 | 11 | 19
  Race: Asian/Oriental | 1 | 1 | 2
  Race: Other | 17 | 22 | 39
  Ethnicity: Hispanic | 73 | 72 | 145
  Ethnicity: Non Hispanic | 85 | 89 | 174
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 8.16 (0.89) | 8.09 (0.96) | 8.12 (0.93)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI was calculated by dividing body weight by the height squared.
  kilogram per square meter (kg/m^2) | 36.76 (7.25) | 36.76 (6.34) | 36.76 (6.80)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 4.40 (3.86) | 4.43 (3.56) | 4.42 (3.70)
Body Weight [Mean (Standard Deviation); unit: kilogram] | 98.51 (23.48) | 100.56 (23.77) | 99.55 (23.61)
2-hour Postprandial Plasma Glucose (PPG) [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] — The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Number of patients analyzed = 158 and 157 for lixisenatide and sitagliptin treatment arm, respectively.
  millimole per liter (mmol/L) | 13.77 (3.78) | 13.92 (3.99) | 13.84 (3.88)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.09 (2.60) | 8.96 (2.59) | 9.03 (2.59)
Glucose Excursion [Mean (Standard Deviation); unit: mmol/L] — Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the meal test, before study drug administration. Number of patients analyzed = 157 and 157 for lixisenatide and sitagliptin treatment arm, respectively.
  mmol/L | 4.37 (2.64) | 4.48 (2.59) | 4.42 (2.61)
Fasting Plasma Insulin (FPI) [Mean (Standard Deviation); unit: picomole/liter (pmol/L)] — Here, number of patients analyzed = 149 and 154 for lixisenatide and sitagliptin treatment arm, respectively.
  picomole/liter (pmol/L) | 108.56 (82.03) | 106.99 (82.69) | 107.76 (82.23)
2-hour Postprandial Plasma Insulin [Mean (Standard Deviation); unit: pmol/L] — Here, number of patients analyzed = 152 and 151 for lixisenatide and sitagliptin treatment arm, respectively.
  pmol/L | 424.67 (350.96) | 420.45 (302.17) | 422.56 (327.02)
Fasting C-Peptide [Mean (Standard Deviation); unit: mmol/L] — Here, number of patients analyzed = 154 and 156 for lixisenatide and sitagliptin treatment arm, respectively.
  mmol/L | 1.19 (0.51) | 1.20 (0.52) | 1.20 (0.52)
2-hour Postprandial C-peptide [Mean (Standard Deviation); unit: mmol/L] — Here, number of patients analyzed = 154 and 156 for lixisenatide and sitagliptin treatment arm, respectively.
  mmol/L | 2.79 (1.28) | 2.92 (1.35) | 2.86 (1.32)
Fasting Glucagon [Mean (Standard Deviation); unit: nanogram/liter (ng/L)] — Here, number of patients analyzed = 154 and 157 for lixisenatide and sitagliptin treatment arm, respectively.
  nanogram/liter (ng/L) | 59.12 (15.81) | 59.43 (20.53) | 59.28 (18.32)
2-hour Postprandial Glucagon [Mean (Standard Deviation); unit: ng/L] — Here, number of patients analyzed = 154 and 155 for lixisenatide and sitagliptin treatment arm, respectively.
  ng/L | 66.36 (17.58) | 67.72 (25.77) | 67.04 (22.05)
Fasting Proinsulin [Mean (Standard Deviation); unit: pmol/L] — Here, number of patients analyzed = 154 and 157 for lixisenatide and sitagliptin treatment arm, respectively.
  pmol/L | 45.06 (39.50) | 44.62 (36.42) | 44.83 (37.91)
2-hour Postprandial Proinsulin [Mean (Standard Deviation); unit: pmol/L] — Here, number of patients analyzed = 154 and 156 for lixisenatide and sitagliptin treatment arm, respectively.
  pmol/L | 105.50 (75.38) | 105.51 (74.00) | 105.51 (74.57)
Fasting Proinsulin-to-Insulin Ratio [Mean (Standard Deviation); unit: ratio] — Here, number of patients analyzed = 149 and 154 for lixisenatide and sitagliptin treatment arm, respectively.
  ratio | 0.53 (0.70) | 0.59 (0.73) | 0.56 (0.71)
2-hour Postprandial Proinsulin-to-Insulin Ratio [Mean (Standard Deviation); unit: ratio] — Here, number of patients analyzed = 152 and 151 for lixisenatide and sitagliptin treatment arm, respectively.
  ratio | 0.36 (0.53) | 0.32 (0.24) | 0.34 (0.41)
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) [Mean (Standard Deviation); unit: milliunit * mmol /liter^2(mU * mmol/L^2)] — HOMA-IR was derived from FPG and FPI as: (FPI [micro units per milliliter] * FPG [mmol/L]) divided by 22.5. Here, number of patients analyzed = 148 and 154 for lixisenatide and sitagliptin treatment arm, respectively.
  milliunit * mmol /liter^2(mU * mmol/L^2) | 6.30 (5.08) | 6.26 (5.32) | 6.28 (5.20)
Homeostatic Model Assessment of Beta-cell Function (HOMA-beta) [Mean (Standard Deviation); unit: percentage of normal beta cells function] — HOMA-beta was derived from FPG and FPI as: (20 * FPI [micro units/milliliter]) divided by (FPG [mmol/L] minus 3.5). Here, number of patients analyzed = 148 and 154 for lixisenatide and sitagliptin treatment arm, respectively.
  percentage of normal beta cells function | 62.01 (59.78) | 60.74 (50.80) | 61.36 (55.29)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than 7% and at Least 5% Weight Loss From Baseline at Week 24
Description: Percentage of patients who met both criteria (HbA1c <7% at Week 24 and at least 5% weight loss from baseline at Week 24) is reported. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Week 24
Population: mITT population included randomized patients who received at least 1 dose of study drug. Missing data was imputed using Last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Groups:
- Lixisenatide: 2-step initiation regimen of lixisenatide along with sitagliptin placebo.
- Sitagliptin: Sitagliptin along with 2-step initiation regimen of volume matching lixisenatide placebo.
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 158 | 161
percentage of participants | 12.0 | 7.5
Statistical Analysis 1: Comparison: Lixisenatide vs Sitagliptin; To demonstrate the superiority of lixisenatide over sitagliptin, 150 patients in each arm would provide a power of 90% with a 2-sided test at the 5% significance level, assuming the percentage of patients defined as responders on HbA1c (<7%) and weight (at least 5% loss) is 25% with lixisenatide and 10% with sitagliptin; Test type: Superiority or Other; p = 0.1696, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel (CMH) test stratified by randomization strata of screening HbA1c (<8.0 or >=8.0%) and randomization strata of screening BMI (<35 or >=35 kg/m^2) was used; Response rate difference = 4.6, 95% CI 2-sided [-1.84 to 11.00], Standard Error of Mean 3.28

2. Secondary Outcome: Absolute Change From Baseline in HbA1c at Week 24
Description: Absolute change = HbA1c value at Week 24 minus HbA1c value at baseline. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed=patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 150 | 160
percentage of hemoglobin | -0.66 (0.094) | -0.72 (0.097)

3. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 152 | 160
kilogram | -2.51 (0.294) | -1.17 (0.304)

4. Secondary Outcome: Change From Baseline in 2-hour Postprandial Plasma Glucose (PPG) at Week 24
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of the study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline 2-hour PPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 129 | 139
mmol/L | -3.35 (0.377) | -1.44 (0.384)

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 1 day after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline FPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 153 | 161
mmol/L | -0.45 (0.193) | -0.69 (0.198)

6. Secondary Outcome: Change From Baseline in Glucose Excursion at Week 24
Description: Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the standardized meal test, before study drug administration. Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of the study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline glucose excursion assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 127 | 139
mmol/L | -2.55 (0.272) | -0.42 (0.275)

7. Secondary Outcome: Change From Baseline in Fasting Plasma Insulin (FPI) and 2-hour Postprandial Plasma Insulin (PPI) at Week 24
Description: Change was calculated for fasting plasma insulin and 2-hour post prandial plasma insulin by subtracting the baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of the study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline plasma insulin assessment during on-treatment period and 'n' = patients with baseline and at least 1 post-baseline assessment for the specified category.
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 123 | 133
pmol/L
  FPI (n=119, 133) | -1.70 (6.789) | -0.88 (7.020)
  2-hour PPI (n=123, 130) | -57.81 (22.788) | -2.85 (23.309)

8. Secondary Outcome: Change From Baseline in Fasting C-peptide and 2-hour Postprandial C-peptide at Week 24
Description: Change was calculated for fasting C-peptide and 2-hour postprandial C-peptide by subtracting the baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline C-peptide assessment during on-treatment period and 'n' = patients with baseline and at least 1 post-baseline assessment for the specified category.
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 125 | 139
nmol/L
  Fasting C-peptide (n= 123,139) | -0.02 (0.039) | -0.02 (0.038)
  2-hour postprandial C-peptide (n=125, 139) | -0.15 (0.100) | 0.08 (0.101)

9. Secondary Outcome: Change From Baseline in Fasting Glucagon and 2-hour Postprandial Glucagon at Week 24
Description: Change was calculated for fasting glucagon and 2-hour postprandial glucagon by subtracting the baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline glucagon assessment during on-treatment period and 'n' = patients with baseline and at least 1 post-baseline assessment for the specified category.
Measure: Least Squares Mean (Standard Error); unit: ng/L
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 124 | 138
ng/L
  Fasting Glucagon (n=124, 138) | 1.89 (1.667) | 3.52 (1.661)
  2-hour postprandial Glucagon (n=124, 134) | -8.16 (1.801) | -4.38 (1.824)

10. Secondary Outcome: Change From Baseline in Fasting Proinsulin and 2-hour Postprandial Proinsulin at Week 24
Description: Change was calculated for fasting proinsulin and 2-hour postprandial proinsulin by subtracting the baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of the study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline proinsulin assessment during on-treatment period and 'n' = patients with baseline and at least 1 post-baseline assessment for the specified category.
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 125 | 140
pmol/L
  Fasting Proinsulin (n=125, 140) | -2.18 (3.172) | -4.84 (3.154)
  2-hour postprandial Proinsulin (n=125, 139) | 0.28 (6.502) | -3.95 (6.477)

11. Secondary Outcome: Change From Baseline in Insulin Resistance Assessed by Homeostasis Model Assessment- Insulin Resistance (HOMA-IR) at Week 24
Description: HOMA-IR was derived from FPG and FPI as: (FPI [micro units per milliliter]*FPG [mmol/L]) divided by 22.5. Change was calculated for HOMA-IR by subtracting the baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HOMA-IR assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mU * mmol/L^2
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 118 | 133
mU * mmol/L^2 | -0.52 (0.366) | -0.57 (0.378)

12. Secondary Outcome: Change From Baseline in Beta Cell Function Assessed by Homeostasis Model Assessment-Beta (HOMA-beta) at Week 24
Description: HOMA-beta was derived from FPG and FPI as: (20*FPI [micro units/milliliter]) divided by (FPG [mmol/L] minus 3.5). Change was calculated for HOMA-beta by subtracting the baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HOMA-beta assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of normal beta cells function
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 118 | 133
percentage of normal beta cells function | 17.66 (9.652) | 17.79 (9.958)

13. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than or Equal to 6.5% at Week 24
Description: The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 150 | 160
percentage of participants | 24.0 | 26.3

14. Other Pre Specified Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than 7% at Week 24
Description: as for outcome 13
Time Frame: Week 24
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 150 | 160
percentage of participants | 40.7 | 40.0

15. Secondary Outcome: Percentage of Patients Requiring Rescue Therapy During 24-Week Period
Description: Routine fasting self-measured plasma glucose (SMPG) and central laboratory FPG (and HbA1c after week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after week 12) were performed. Threshold values - from baseline to Week 8: fasting SMPG/FPG >270 milligram/deciliter (mg/dL) (15.0 mmol/L), from Week 8 to Week 12: fasting SMPG/FPG >240 mg/dL (13.3 mmol/L), and from Week 12 to Week 24: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c >8.5%.
Time Frame: Baseline up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 158 | 161
percentage of participants | 9.5 | 6.8

16. Other Pre Specified Outcome: Percentage of Patients With at Least 5% Weight Loss From Baseline at Week 24
Description: as for outcome 13
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 152 | 160
percentage of participants | 18.4 | 11.9

17. Other Pre Specified Outcome: Change From Baseline in Fasting Proinsulin-to-insulin Ratio and 2-hour Postprandial Proinsulin-to-insulin Ratio at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of the study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline proinsulin-to-insulin ratio assessment during on-treatment period and 'n' = patients with baseline and at least 1 post-baseline assessment for the specified category.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 123 | 133
ratio
  Fasting Proinsulin-to-insulin ratio (n=119, 133) | -0.08 (0.035) | -0.17 (0.036)
  2-hour PP Proinsulin-to-insulin ratio (n=123, 130) | -0.01 (0.025) | -0.05 (0.026)

18. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia and Severe Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the patient required the assistance of another person and was associated with either a plasma glucose level below 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose administration
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lixisenatide | Sitagliptin
Number analyzed (Participants) | 158 | 161
participants
  Symptomatic hypoglycemia | 1 | 3
  Severe symptomatic hypoglycemia | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 3 days after the last dose administration
Description: Median exposure to study treatment was 169.0 days in both lixisenatide and sitagliptin treatment arm. The analysis was performed on safety population, defined as all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Arm/Group | Lixisenatide | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 3/158 | 3/161
Other Adverse Events (participants affected / at risk) | 54/158 | 45/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide (N=158) | Sitagliptin (N=161)
Abscess limb (Infections and infestations) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide (N=158) | Sitagliptin (N=161)
Influenza (Infections and infestations) | 8 | 5
Nasopharyngitis (Infections and infestations) | 10 | 12
Dizziness (Nervous system disorders) | 8 | 5
Headache (Nervous system disorders) | 20 | 15
Diarrhoea (Gastrointestinal disorders) | 14 | 12
Nausea (Gastrointestinal disorders) | 28 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.